CLINICAL TRIAL: NCT03356210
Title: Quantitative Electroencephalography and Neurofeedback Training for the Treatment of Substance Use Disorders: A Randomized Controlled Trial
Brief Title: Neurofeedback Training for the Treatment of Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSHF_2017
Record Dates: First submitted 2017-07-14; First posted 2017-11-29 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2020-01

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants doing follow-up assessment will be blinded to condition assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (No Intervention): This control group will receive treatment as usual; conventional counseling
- Neurofeedback + TAU (Experimental): 20 sessions of symptom-based NF training in conjunction with traditional therapy
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback — The intervention will consist of 20 sessions of symptom-based NF tailored to the individual patient. Training will be conducted using the Othmer method of NF from EEGinfo, comprising bipolar, infra-low frequency training, with the inclusion of synchrony and alfa-/theta training as needed.
  Arms: Neurofeedback + TAU

SUMMARY:
The proposed randomized controlled trial (RCT) will investigate the usefulness of electroencephalographic (EEG) biofeedback, also called neurofeedback (NF), a treatment method that can potentially prevent relapses among patients with a substance use disorder (SUD) through its calming effect on the central nervous system.

The study will examine whether NF can improve general well-being and quality of life (QoL) and subsequently its ability to play a role in relapse prevention strategies. Specifically, the effect on physical and psychological distress will be investigated.

DETAILED DESCRIPTION:
A patient with a substance use disorder (SUD) typically requires comprehensive and individualized care across different levels of service providers, from primary care to the specialist health care services. Among the known threats to a prolonged remission are negative emotional states because they can trigger the urge to use drugs. An integrative approach is warranted aimed to address the physiological, psychological and social aspects of the disorder during the rehabilitation period.

Patients with a SUD diagnosis in an outpatient clinic will be randomized to either 1) 20 sessions of symptom-based NF training in conjunction with traditional therapy or 2) conventional counseling. The primary outcome is QoL at the end of treatment and at a 3 and 12 month follow-up. Secondary outcome measures include alcohol and drug use, mental distress, sleep quality and cognitive function. The optimal quantity of the intervention will be assessed with a cost-benefit approach.

The proposed study will provide new knowledge about how NF can be best utilized in SUD treatment, potentially improving QoL and relapse rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a substance use disorder referred to outpatient addiction treatment, aged >18 of both genders.

Exclusion Criteria:

* Severe psychiatric disorders (e.g. psychosis) that have not been stabilized with e.g., medication (assessed as a part of the clinical process at the clinic). Severe cognitive impairment or language problems (inability to converse for interviews).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) | After the intervention (approx 5 months)
  QoL is measured with the Quality of Life 5 scale (QoL-5). QoL-5 consists of five subjective statements: two questions are about health, physical and mental; two questions address the quality of significant relationships (partner and friends); and one question addresses the existential self i.e. the relationship with oneself. Responses are scored on a 5-step ordinal scale from 1 to 5. A score of 1 is very good, and 5, very poor. The scores are transposed, and inverted into a decimal scale ranging from 0.1 to 0.9; 0.9 is now the best score and 0.1, the worst. Mean scores for health and relationship QoL are calculated, and a total QoL score is calculated as a mean of health, relationship and existential QoL.
Quality of life at 3 months follow up | Short term outcome - 3 months follow-up
  QoL is measured with the Quality of Life 5 scale (QoL-5). QoL-5 consists of five subjective statements: two questions are about health, physical and mental; two questions address the quality of significant relationships (partner and friends); and one question addresses the existential self i.e. the relationship with oneself. Responses are scored on a 5-step ordinal scale from 1 to 5. A score of 1 is very good, and 5, very poor. The scores are transposed, and inverted into a decimal scale ranging from 0.1 to 0.9; 0.9 is now the best score and 0.1, the worst. Mean scores for health and relationship QoL are calculated, and a total QoL score is calculated as a mean of health, relationship and existential QoL.
Quality of life at 12 months follow-up | Long-term outcome - 12 months follow-up
  QoL is measured with the Quality of Life 5 scale (QoL-5). QoL-5 consists of five subjective statements: two questions are about health, physical and mental; two questions address the quality of significant relationships (partner and friends); and one question addresses the existential self i.e. the relationship with oneself. Responses are scored on a 5-step ordinal scale from 1 to 5. A score of 1 is very good, and 5, very poor. The scores are transposed, and inverted into a decimal scale ranging from 0.1 to 0.9; 0.9 is now the best score and 0.1, the worst. Mean scores for health and relationship QoL are calculated, and a total QoL score is calculated as a mean of health, relationship and existential QoL. Normative data from a previous survey of the general population showed a mean QoL score of 0.69 and a minimal clinically important difference is 0.10.

SECONDARY OUTCOMES:
Perceived functioning/well-being | After the intervention (approx 5 months) and 3 & 12 months follow-up
  Perceived functioning/well-being will be measured with the Outcome rating scale (ORS). The ORS each consist of four 10-cm visual analog scales (VAS) ranging from negative (left) to positive (right). The ORS measures three areas of client functioning: individual, interpersonal, and social, as well as measuring the client's overall view of their personal well-being. The marks made by clients on each of the four lines are measured to the nearest millimeter to derive the score. These are then summed to obtain a total score. Cm is analogue to scale score and the total score range from 0 to 40. High scores reflect a good level of well-being and functioning. A clinical cut-off is 25 (i.e., one would expect scores below 25 in a clinical sample) and a 5 point difference in score is consider as the minimal clinically important difference
Perceived psychological distress | After the intervention (approx 5 months) and 3 & 12 months follow-up
  Perceived psychological distress measured with the Symptom Check List - 10 (SCL-10), a short-form of the Hopkins Symptom Checklist 90. SCL-10 has 10 items about anxiety (4 items) and depression (6 items). Responses are scored on an ordinal scale from 1 to 4, with the highest score indicating highest distress. A total mean score is calculated. Scores above 1.85 is considered a pathological score.
Substance use | After the intervention (approx 5 months) and 3 & 12 months follow-up
  Substance use will be assessed with the European version of the Addiction Severity index (EuropASI). Data on drug and alcohol use in the 30 days before the interview are used to derive a composite score to indicate severity; scores range from 0 (no problem) to 1 (a severe problem).
Physiological variables | After the intervention (approx 5 months) and 3 & 12 months follow-up
  Sleep quality will be assessed using a 10-cm visual analog scale (VAS) ranging from negative (left) to positive (right).
Drop-out | After the intervention (approx 5 months) and 3 & 12 months follow-up
  Drop-out rates from the out-patient treatment, i.e., the percentage who has dropped-out of treatment in each group.
Restlessness & trepidation | After the intervention (approx 5 months) and 3 & 12 months follow-up
  Restlessness & trepidation will be assessed using a 10-cm visual analog scales (VAS) ranging from negative (left) to positive (right).

CONTACTS AND LOCATIONS:
Overall Officials: John-Kåre Vederhus, PhD, Principal Investigator — Addiction Unit, Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital HF, Kristiansand, Vest Agder, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymized after study completion and will then be deposited to the publicly available data repository of the Norwegian Centre for Research Data.
Supporting Information: Study Protocol, ICF
Time Frame: After study completion and writing up of results, expected 31.12.22
Access Criteria: Open

REFERENCES:
- [Derived] Gabrielsen KB, Clausen T, Haugland SH, Hollup SA, Vederhus JK. Infralow neurofeedback in the treatment of substance use disorders: a randomized controlled trial. J Psychiatry Neurosci. 2022 Jun 15;47(3):E222-E229. doi: 10.1503/jpn.210202. Print 2022 May-Jun. PMID 35705204

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03356210/Prot_SAP_000.pdf